CLINICAL TRIAL: NCT03486704
Title: The Italian Network of Telerehabilitation: Evaluation of Telerehabilitation System in Mild Cognitive Impairment
Brief Title: Telerehabilitation in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: IRCCS Centro Neurolesi Bonino Pulejo (Other); Fondazione Don Carlo Gnocchi Onlus (Other); IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR-Rehab-MCI
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-03

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Face to Face VRRS and telerehabilitation (Experimental): Participants will receive 12 sessions of an individualized Face to Face cognitive training using VRRS over 4 weeks followed by 36 sessions of home-based VRRS cognitive training, three sessions for week.
  Interventions: Behavioral: Face to Face VRRS and telerehabilitation
- Usual rehabilitation program (Active Comparator): The usual rehabilitation group will receive 12 sessions of face-to-face usual cognitive training program.
  Interventions: Behavioral: Usual rehabilitation program
- FTF VRRS plus unstructured CS (Active Comparator): Participants will receive 12 sessions of an individualized Face to Face (FTF) cognitive training using VRRS over 4 weeks followed by 36 sessions of home-based unstructured cognitive stimulation (CS), three sessions for week.
  Interventions: Behavioral: FTF VRRS plus unstructured CS
- Face to Face VRRS plus active tDCS and telerehabilitation (Experimental): Participants will receive 12 sessions of an individualized Face to Face cognitive training using VRRS combined with active (anodal) tDCS applied to the left dorsolateral prefrontal cortex over 4 weeks followed by 36 sessions of home-based VRRS cognitive training, three sessions for week.
  Interventions: Behavioral: Face to Face VRRS plus active tDCS and telerehabilitation
- Face to Face VRRS plus placebo tDCS and telerehabilitation (Active Comparator): Participants will receive 12 sessions of an individualized Face to Face cognitive training using VRRS combined with placebo tDCS applied to the dorsolateral prefrontal cortex of the left hemisphere over 4 weeks followed by 36 sessions of home-based VRRS cognitive training, three sessions for week.
  Interventions: Behavioral: Face to Face VRRS plus placebo tDCS and telerehabilitation

INTERVENTIONS:
Behavioral: Face to Face VRRS and telerehabilitation — Face to Face cognitive training using VRRS plus telerehabilitation. Participants will receive 12 sessions of an individualized Face to Face cognitive training using VRRS over 4 weeks followed by 36 sessions of home-based VRRS cognitive training, three sessions for week.
  Cognitive training will initially be tailored to the patient's baseline characteristics. The exercise program will be charged by therapist on the patient's computer before the beginning of the at-home treatment. Each patient's performed session will be reviewed by the therapist.
  The group will receive a kit home-based (a tablet home, access to a daily individualized cognitive training program).
  Arms: Face to Face VRRS and telerehabilitation
Behavioral: Usual rehabilitation program — The usual rehabilitation group will receive 12 sessions of face-to-face usual cognitive training program.
  Arms: Usual rehabilitation program
Behavioral: FTF VRRS plus unstructured CS — Face to Face cognitive training using VRRS plus at-home unstructured cognitive stimulation.
  Participants will receive 12 sessions of an individualized Face to Face (FTF) cognitive training using VRRS over 4 weeks followed by 36 sessions of home-based unstructured cognitive stimulation (CS), three sessions for week.
  Arms: FTF VRRS plus unstructured CS
Behavioral: Face to Face VRRS plus active tDCS and telerehabilitation — Participants will receive 12 sessions of an individualized Face to Face cognitive training using VRRS combined with active (anodal) tDCS applied to the left dorsolateral prefrontal cortex over 4 weeks followed by 36 sessions of home-based VRRS cognitive training, three sessions for week.
  Face to Face VRRS cognitive training will initially be tailored to the patient's baseline characteristics.
  The exercise program will be charged by therapist on the patient's computer before the beginning of the at-home treatment. Each patient's performed session will be reviewed by the therapist.The group will receive a kit home-based (a tablet home, access to a daily individualized cognitive training program).
  Arms: Face to Face VRRS plus active tDCS and telerehabilitation
Behavioral: Face to Face VRRS plus placebo tDCS and telerehabilitation — Participants will receive 12 sessions of an individualized Face to Face cognitive training using VRRS combined with placebo tDCS applied to the dorsolateral prefrontal cortex of the left hemisphere over 4 weeks followed by 36 sessions of home-based VRRS cognitive training, three sessions for week.
  Face to Face VRRS cognitive training will initially be tailored to the patient's baseline characteristics.
  The exercise program will be charged by therapist on the patient's computer before the beginning of the at-home treatment. Each patient's performed session will be reviewed by the therapist.The group will receive a kit home-based (a tablet home, access to a daily individualized cognitive training program).
  Arms: Face to Face VRRS plus placebo tDCS and telerehabilitation

SUMMARY:
The main aim of the study is to evaluate the efficacy of the Virtual Reality Rehabilitation System (VRRS) compared to usual care treatment for patients with Mild Cognitive Impairment (MCI). Moreover, we will assess the possibility to prolong the beneficial effects of the treatment with an innovative telerehabilitation system. In the second phase of the present study we aim to evaluate the short and long term effects induced by the treatment of active (anodal) transcranial Direct Current Stimulation (tDCS) applied to the left dorsolateral prefrontal cortex combined with VRRS compared to placebo tDCS stimulation combined with VRRS.

The effects of the intervention on outcome variables will be assessed using a randomized controlled trial design with five groups. The investigators will assess the effects of VRRS system and of the implementation of the at-home treatment on the quality of life, cognitive and functional abilities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MCI, defined according to standard criteria (Petersen et al., 2011)
* Mini Mental State Examination (MMSE) ≥24
* Education ≥ 5 years
* All of the subjects will have normal or corrected-to-normal vision and will be native Italian speakers.
* All participants reported subjective memory complaints and objective memory impairment, but no impairment of function in daily life.

Exclusion Criteria:

* visual perception disorder and/or hearing loss
* history of major psychiatric disorders
* any contraindication for tDCS such as a history of seizures, major head trauma, past brain surgery, a brain metal implant or a pacemaker.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in long term episodic verbal memory | Baseline up to 12 weeks and 4 and 7 months
  Free and Cued Selective Reminding Test (FCSRT)
Change in long term episodic verbal memory | Baseline up to 12 weeks and 4 and 7 months
  Auditory Verbal Learning Test, immediate and delayed recall

SECONDARY OUTCOMES:
Change in measure of quality of life | Baseline up to 12 weeks and 4 and 7 months
  Quality of Life in Alzheimer's Disease (AD) - QoL-AD
Change in dementia severity | Baseline up to 12 weeks and 4 and 7 months
  Clinical Dementia Rating scale (CDR)
Change in global cognition | Baseline up to 12 weeks and 4 and 7 months
  Mini Mental State Examination (MMSE)
Change in memory complaints | Baseline up to 12 weeks and 4 and 7 months
  Everyday Memory Questionnaire (EMQ)
Change in visual constructional abilities | Baseline up to 12 weeks and 4 and 7 months
  Rey-Osterrieth Figure Copy
Change in nonverbal long term memory | Baseline up to 12 weeks and 4 and 7 months
  Rey-Osterrieth Figure Recall
Change in visual attention and task switching | Baseline up to 12 weeks and 4 and 7 months
  Trail Making Test
Change in naming abilities | Baseline up to 12 weeks and 4 and 7 months
  Object and action naming subtests of the Battery for the Analysis of the Aphasic Deficit
Change in non-verbal abstract reasoning | Baseline up to 12 weeks and 4 and 7 months
  Raven's Colored Progressive Matrices
Change in verbal fluency | Baseline up to 12 weeks and 4 and 7 months
  Phonemic verbal fluency and semantic verbal fluency

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro san Giovanni di Dio, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manenti R, Baglio F, Pagnoni I, Gobbi E, Campana E, Alaimo C, Rossetto F, Di Tella S, Pagliari C, Geviti A, Bonfiglio NS, Calabro RS, Cimino V, Binetti G, Quartarone A, Bramanti P, Cappa SF, Rossini PM, Cotelli M. Long-lasting improvements in episodic memory among subjects with mild cognitive impairment who received transcranial direct current stimulation combined with cognitive treatment and telerehabilitation: a multicentre, randomized, active-controlled study. Front Aging Neurosci. 2024 Jun 18;16:1414593. doi: 10.3389/fnagi.2024.1414593. eCollection 2024. PMID 38966802
- [Derived] Manenti R, Gobbi E, Baglio F, Macis A, Ferrari C, Pagnoni I, Rossetto F, Di Tella S, Alemanno F, Cimino V, Binetti G, Iannaccone S, Bramanti P, Cappa SF, Cotelli M. Effectiveness of an Innovative Cognitive Treatment and Telerehabilitation on Subjects With Mild Cognitive Impairment: A Multicenter, Randomized, Active-Controlled Study. Front Aging Neurosci. 2020 Nov 16;12:585988. doi: 10.3389/fnagi.2020.585988. eCollection 2020. PMID 33304267